CLINICAL TRIAL: NCT03258671
Title: IMRT and Timing in Combination With EGFRTKI for Stage IV Non-small-cell Lung Cancer: Results of a Randomised,Openlabel,Multicentre Study
Brief Title: IMRT and Timing in Combination With EGFRTKI for Stage IV Non-small-cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LuBing (Other)
Responsible Party: Sponsor-Investigator, LuBing, Director, Guizhou Medical University
Organization: Guizhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSWOG
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Non-Small Cell Lung Cancer; Nonsmall Cell Lung Cancer; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mutation+ concurrent (Experimental): IMRT concurrent with EGFR-TKI on paticipants with known sensitive EGFR mutations.
  Interventions: Drug: EGFR-TK Inhibitor; Radiation: Intensity Modulated Radiation Therapy
- Mutation+ concomitant (Experimental): IMRT concomitant with EGFR-TKI on paticipants with known sensitive EGFR mutations.
  Interventions: Drug: EGFR-TK Inhibitor; Radiation: Intensity Modulated Radiation Therapy

INTERVENTIONS:
Drug: EGFR-TK Inhibitor — ·EGFR-TKI：gefitinib will be administered 250mg/d ivgtt qd; icotinib will be administered 150mg/d ivgtt tid;
Radiation: Intensity Modulated Radiation Therapy — High dose group：DTGTV=70Gy；
  * first course radiotherapy：40Gy/20f/4w（DTPTV：36Gy/20f/4w）,2Gy/f/d；
  * late course radiotherapy：1.5Gy/f、2f/d、interval≥6 hs、DTGTV=30Gy（DTPTV=27Gy）。
  Low dose group：DTGTV=50Gy;
  * first course radiotherapy：32Gy/16f/3w（DTPTV为28.8Gy/16f/3w），2Gy/f/d；
  * late course radiotherapy：1.5Gy/f、2f/d、interval≥6小时、DTGTV为18Gy（DTPTV为16.2Gy）。

SUMMARY:
This study is for patients with EFGR gene sensitive mutations diagnosed by pathology or cytology, having a course of chest radiotherapy treatment and molecular Target Therapy for the treatment of stage IV non-small cell lung cancer. Patients with non-small cell lung cancer have a risk of the tumour in the lung recurring or progressing after treatment.

In this study, the investigators aim to verify the following hypothesis:

* whether in combination with concurrent or concomitant EGFR-TKI regimen chemotherapy, Intensity Modulated Radiation Therapy can reduce the risk of the tumour in the lung recurring or progressing similarily.
* Intensity Modulated Radiation Therapy concomitant with EGFR-TKI has a better normal tissue dose/volume tolerance than concurrent regimen.
* the survival can be improved by using this new molecular Target-radiotherapy method.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IV NSCLC[UICC 2017 8th edition] with known sensitive EGFR mutations(confirmed by tissue or blood).
* Have not received one or more prior treatments
* 18 to 80 years of age.ECOG performance status 0～2 or KPS≥60
* Have distant metastatic lesions≤5；and have clear consciousness when the metastatic sites were brain; and have no influence on pulmonary function when the metastatic sites were lung.
* Have no contraindications in radiotherapy, EGFR-TKI and chemotherapy
* Normal bone marrow and organ function as defined below:

Absolute neutrophil count ≥ 1,500/mcl Platelets ≥ 100,000/mcl Hemoglobin ≥ 9.0 g/dL Total bilirubin ≤ 2.0 x IULN AST (SGOT) / ALT (SGPT) ≤ 3.0 x IULN; if liver metastases, ≤ 5.0 x IULN Serum creatinine ≤ 1.5 x ULN LVEF ≥ 50% performed no more than 4 weeks prior to enrollment. FEV1>50%，mild-moderate pulmonary function dysfunction.

* Able to understand and willing to sign a Human Research Protection Office (HRPO) approved written informed consent document (or that of legally authorized representative, if applicable).
* With good compliance to the treatment and Follow-up

Exclusion Criteria:

* Evidence of small cell, large cell neuroendocrine or carcinoid histology.
* Non-stage IV NSCLC and ECOG performance status 3～5 or KPS<60
* Have a serious or uncontrolled medical condition that could compromise the patients' ability to adhere to the protocol.
* Malignant pleural effusion and pericardial effusion
* Uncontrolled intercurrent illness including, but not limited to, hypertension , diabetes mellitus ,ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding: Patient must have a negative pregnancy test within 14 days of study entry.
* Have a secondary malignancy (except adequately treated non-melanomatous skin cancer, or other cancer such as in situ of the cervix. considered cured by surgical resection or radiation). Patients who have had another malignancy in the past but have been disease free for more than 5 years are eligible.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to EGFR-TKI or other agents used in the study.
* With poor compliance
* The researchers consider it inappropriate to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Therapeutic efficacy of EGFR-TKI and concurrent/concomitant local RT in NSCLC patients. | >4 weeks post treatment
  Tumor Response will be evaluated using the RECIST system. Modified WHO criteria will be used for measurement of tumors. The irradiated lesion will be excluded from the assessment of response.
Overall survival (OS) | Up to 5 years
  Overall survival is defined as the time interval from date of diagnosis to date of death from any cause
Progression-free survival (PFS) | Up to 5 years
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  Progressive disease (PD) = at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, appearance of one or more non-target lesion(s) and/or unequivocal progression of existing non-target lesions

SECONDARY OUTCOMES:
Objective response rate(ORR) | Up to 5 years
  Partial response + complete response per RECIST 1.1 criteria Complete response (CR) = disappearance of all target lesions, non-target lesions, and normalization of tumor marker level
  Partial response (PR) = at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline of sum diameters
Disease control rate (DCR) | Up to 5 years
  Percentage of patients who achieve complete response, partial response, or stable disease per RECIST 1.1 criteria.
  Complete response (CR) = disappearance of all target lesions, non-target lesions, and normalization of tumor marker level
  Partial response (PR) = at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline of sum diameters
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Adverse events (toxicities) | Up to 5 years
  The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Local regional progression-free survival（LRPFS） | Time Frame: Up to 5 years
  LRPFS is defined as the duration of time from start of treatment to time of progression or recurrence, whichever occurs first..The target lesions is only for primary tumor and regional positive lymph nodes.
  Progressive disease (PD) = at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, appearance of one or more target lesion(s) and/or unequivocal progression of existing target lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Bing, Director, Study Director — ouyangww103173@163.com
Locations (1):
- The affiliated hospital of Guizhou medical university, Guiyang, Guizhou, China

REFERENCES:
- [Derived] Li Q, Liang N, Zhang X, Zhang Y, Ouyang W, Su S, Ma Z, Hu Y, Geng Y, Chen X, Lu B. Reasonable Timing of Radiotherapy for Stage IV Non-Small-Cell Lung Cancer During Targeted Therapy Based on Tumour Volume Change. Front Oncol. 2021 Sep 23;11:705303. doi: 10.3389/fonc.2021.705303. eCollection 2021. PMID 34631535